CLINICAL TRIAL: NCT05026450
Title: Exploring the Psycho-traumatic Impact of a Violent Act Commited - Study Among Inmates of the Bordeaux-Gradignan Penitentiary Center
Brief Title: Exploring the Psycho-traumatic Impact of a Violent Act Commited at the Bordeaux-Gradignan Penitentiary Center
Acronym: IPTAVC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Charles Perrens, Bordeaux (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-A01298-33
Record Dates: First submitted 2021-08-17; First posted 2021-08-30 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Post Traumatic Stress Disorder; Offensive Aggression; Violent Behavior
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will seek to explore the possibility of developing post-traumatic stress disorder following a violent offense commited, among the population of prisoners of the Bordeaux-Gradignan penitentiary center.

DETAILED DESCRIPTION:
The overrepresentation of psychiatric disorders among prisoners has been the subject of numerous studies and the significant increase in the number of prisoners over the past 3 decades, make research in prisons a major public health issue.

Recent studies have been able to highlight an over-representation of post-traumatic stress disorder in the prison population. Leading to questionning the factors that could explain the overrepresentation of this disorder in prison with various hypotheses raised. Among these hypotheses, the possibility of developing post-traumatic stress disorder following a violent offense commited has been proposed.

The study will thus seek to explore the development of a Post-traumatic Stress Disorder following a violent act committed using the PCL-5 questionnaire

Study design :Observational, descriptive, monocentric study with completion of an anonymous self-questionnaire.

Participation in the study is voluntary and anonymous with signature of a non-opposition form.

Expected outcomes : better knowledge of this disorder in detention and a hypothesis to explain its overrepresentation. Earlier detection of this pathology in prison could thus be considered, in particular by improving the identification of people at risk according to the presence of contributing factors. More specific support and improved access to care for inmates could be considered, allowing early treatment and thus avoiding progression to other co-morbidities or risk of recidivism.

ELIGIBILITY:
Inclusion Criteria

* Aged over 18
* Have as a reason for imprisonment one of the following: Homicide and willful violence resulting in death, Rape or sexual assault, Violence and other personal injury.
* Having signed and duly completed the Non-Objection form for participation in the study
* Mastery of the French language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prisoners incarcerated in the Bordeaux-Gradignan penitentiary center.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Explore whether Post-Traumatic Stress Disorder develops as a result of a violent act committed. | 1 month
  Evaluation of Post-traumatic stress disorder using the PTSD self-report scale: PCL-5, with a cut-off value of 38 to indicate the presence of a diagnosis of PTSD.

SECONDARY OUTCOMES:
Identify risk factors that may have contributed to the onset of symptoms of post-traumatic stress disorder | Baseline
  Socio-demographic data, personnal and medical history
Identify risk factors that may have contributed to the maintenance of symptoms of post-traumatic stress disorder | 1 month
  Socio-demographic data, personnal and medical history
Frequency of post-traumatic stress disorder according to the various factors that may have contributed to its onset | 1 month
  Age, sex, length of time since the offense, possible link with the victim, history of psychiatric follow-up and history of exposure to other traumatic events

CONTACTS AND LOCATIONS:
Overall Officials: Severine BEAUVAIS, MD, Principal Investigator — CH CharlesPerrens
Locations (1):
- Centre Hospitalier Charles PERRENS, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No
no IPD sharing plan

REFERENCES:
- [Background] Koenen KC, Ratanatharathorn A, Ng L, McLaughlin KA, Bromet EJ, Stein DJ, Karam EG, Meron Ruscio A, Benjet C, Scott K, Atwoli L, Petukhova M, Lim CCW, Aguilar-Gaxiola S, Al-Hamzawi A, Alonso J, Bunting B, Ciutan M, de Girolamo G, Degenhardt L, Gureje O, Haro JM, Huang Y, Kawakami N, Lee S, Navarro-Mateu F, Pennell BE, Piazza M, Sampson N, Ten Have M, Torres Y, Viana MC, Williams D, Xavier M, Kessler RC. Posttraumatic stress disorder in the World Mental Health Surveys. Psychol Med. 2017 Oct;47(13):2260-2274. doi: 10.1017/S0033291717000708. Epub 2017 Apr 7. PMID 28385165
- [Background] Baranyi G, Cassidy M, Fazel S, Priebe S, Mundt AP. Prevalence of Posttraumatic Stress Disorder in Prisoners. Epidemiol Rev. 2018 Jun 1;40(1):134-145. doi: 10.1093/epirev/mxx015. PMID 29596582
- [Background] Fazel S, Baillargeon J. The health of prisoners. Lancet. 2011 Mar 12;377(9769):956-65. doi: 10.1016/S0140-6736(10)61053-7. Epub 2010 Nov 18. PMID 21093904
- [Background] Ashbaugh AR, Houle-Johnson S, Herbert C, El-Hage W, Brunet A. Psychometric Validation of the English and French Versions of the Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5). PLoS One. 2016 Oct 10;11(10):e0161645. doi: 10.1371/journal.pone.0161645. eCollection 2016. PMID 27723815
- [Background] Jakobowitz S, Bebbington P, McKenzie N, Iveson R, Duffield G, Kerr M, Killaspy H. Assessing needs for psychiatric treatment in prisoners: 2. Met and unmet need. Soc Psychiatry Psychiatr Epidemiol. 2017 Feb;52(2):231-240. doi: 10.1007/s00127-016-1313-5. Epub 2016 Nov 22. PMID 27878323
- [Background] Vaiva G, Jehel L, Cottencin O, Ducrocq F, Duchet C, Omnes C, Genest P, Rouillon F, Roelandt JL. [Prevalence of trauma-related disorders in the French WHO study: Sante mentale en population generale (SMPG)]. Encephale. 2008 Dec;34(6):577-83. doi: 10.1016/j.encep.2007.11.006. Epub 2008 Apr 2. French. PMID 19081454